CLINICAL TRIAL: NCT02054182
Title: Effect of Vitamin D Supplementation in Young Children With Acute Lower Respiratory Tract Infection at Dr George Mukhari Academic Hospital, Pretoria, South Africa
Brief Title: Effect of Vitamin D Supplementation in Young South African Children Hospitalized With Acute Lower Respiratory Infection
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Limpopo (Other)
Responsible Party: Principal Investigator, Siyazi Mda, Research project supervisor, University of Limpopo
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MREC/M/83/2013:PG
Record Dates: First submitted 2014-01-18; First posted 2014-02-04 (Estimated); Last update posted 2014-02-04 (Estimated); Status verified 2014-01

CONDITIONS: Acute Lower Respiratory Tract Infection; Pneumonia; Bronchiolitis
Keywords: vitamin D supplementation, pneumonia, bronchiolitis
MeSH Terms: conditions — Pneumonia; Bronchiolitis | interventions — Vitamin D; Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vitamin D (Active Comparator): Vitamin D 2 500 IU daily from enrolment until hospital discharge
  Interventions: Drug: Vitamin D
- Placebo (Placebo Comparator): Placebo

INTERVENTIONS:
Drug: Vitamin D — Vitamin D 2 500 IU daily from enrolment (within 24 hours of hospitalization) until discharge from hospital
  Other Names: Cholecalciferol
  Arms: Vitamin D

SUMMARY:
The purpose of this study is to determine whether vitamin D supplements given to children aged 1 month to 5 years, hospitalized with acute lower respiratory tract infection will improve symptoms and reduce the duration of hospitalization.

DETAILED DESCRIPTION:
In a randomized, double blind placebo controlled interventional study, children aged 1 month to 5 years, who are admitted with acute lower respiratory tract infection (ALRTI) to Dr George Mukhari Academic Hospital will be enrolled. The children will randomized to receive 2500 IU of vitamin D or a placebo. It is intended to enrol 320 children, 160 to receive vitamin D and the other 160 to receive a placebo. This sample size was calculated at 80% power and 5% significance. The children will be enrolled within 24 hours of admission and the intervention (supplement or placebo) will be daily until the child is discharged fron the hospital.

The severity of ALRTI will be assessed using the modified Respiratory Distress Assessment Instrument (MRDAI) score. The thorough physical examination and classification of severity of the symptoms will be done at enrolment and daily until hospital discharge.

Blood samples for vitamin D and calcium concentrations will be assessed at enrolment, before the child is given the supplement or placebo.

The difference in the improvement in MRDAI score between the placebo and the supplement will be assessed by analysis of variance (ANOVA). Similarly the difference in duration of hospital stay between the two groups will also be analysed using ANOVA. The association between the vitamin D levels and the MRDAI score on admission will also be assessed and analysed using ANOVA.

All eligible children will be sequentially enrolled until the desired sample size is reached. A simple randomisation by means of computer generated numbers will be used to minimize selection bias. Both the study subjects and the investigators will be blinded to the allocation (treatment or placebo). The unblinding will be done only after the analysis has been completed.

ELIGIBILITY:
Inclusion Criteria:

* All children age 1month - 5 yrs, admitted in the paediatric unit of Dr George Mukhari Hospital with an acute lower respiratory tract infection i.e. bronchiolitis and/ or pneumonia

Exclusion Criteria:

* Children whose caregivers decline participation in the study Children with co-morbid chronic respiratory condition(s) Children who have received vitamin D supplementation in the past 30 days

Ages: 1 Month to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 320 (Estimated)
Dates: Start 2014-02; Primary Completion 2014-11 (Estimated); Study Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
Comparison of change from baseline in modified Respiratory Distress Assessment Instrument score at hospital discharge between vitamin D supplement and placebo groups. | Participants will be followed for the duration of hospital stay, an expected average of 7 days
  The modified Respiratory Distress Assessment Instrument score, involves the measurement of the child's respiratory rate, assessment of the use of accessory muscles, the child's color, and auscultatory findings; each of these is given a score from 0 to 3. The higher the score the more severe the clinical condition. This scoring system has been validated in a number of scientific studies.

SECONDARY OUTCOMES:
Comparison of duration of hospitalization between vitamin D supplementation and placebo groups. | Participants will be followed for the duration of hospital stay, an expected average of 7 days
  The duration of hospital stay will be calculated from the day of admission to the day the child is assessed and deemed fit for discharge by the attending physician. All children at discharge will have a modified RDAI score of less than 3.

OTHER OUTCOMES:
Assessment of correlation between vitamin D levels and modified Respiratory Distress Assessment Instrument score | On day 1, i.e. date of randomization
  Blood for vitamin D levels will be obtained at enrolment and this will be used to assess whether a child is vitamin D deficient. Severity of ALRTI symptoms will also be assessed at enrolment using the modified RDAI. The correlation between vitamin D deficiency and severity of symptoms will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Siyazi Mda, MBChB, PhD, Study Chair — Univeristy of Limpopo, Medunsa Campus
Locations (1):
- Dr George Mukhari Academic Hospital, Pretoria, Gauteng, South Africa